CLINICAL TRIAL: NCT06107907
Title: Using Electrical Impedance Tomography to Investigate the Relationship Between Airflow Rate During High-flow Oxygen Therapy and Pressure in Patients With Heart Failure Compared to Non-invasive Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202307158DINA
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: to Assess the Corresponding PEEP Values in NIV With CPAP Under Different Airflow Rates During HFOT in Heart Failure Patients
Keywords: Electrical Impedance Tomography; non-invasive ventilator; high flow oxygen therapy; Positive end-expiratory pressure; Continuous positive airway pressure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): follow the sequence of oxygen mask, HFOT 40L, HFOT 50L, HFOT 60L, oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, and CPAP 6cmH2O.
  Interventions: Device: Non-invasive ventilation (NIV) or high-flow oxygen therapy (HFOT) using electrical impedance tomography (EIT)
- Group B (Other): follow the sequence of oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, CPAP 6cmH2O, oxygen mask, HFOT 40L, HFOT 50L, and HFOT 60L.
  Interventions: Device: Non-invasive ventilation (NIV) or high-flow oxygen therapy (HFOT) using electrical impedance tomography (EIT)

INTERVENTIONS:
Device: Non-invasive ventilation (NIV) or high-flow oxygen therapy (HFOT) using electrical impedance tomography (EIT) — Participants will be randomly assigned to Groups A and B using a computerized randomization process. Each group will undergo specific protocols for 5-10 minutes per phase. NIV will be administered in continuous positive airway pressure (CPAP) mode. The participants will be positioned in a semi-recumbent position at 45 degrees, and the EIT belt will be placed around the fifth (or sixth) intercostal space for monitoring. The EIT signals will be filtered with a cut-off frequency set at 10 beats below the current heart rate. The entire procedure is estimated to take approximately 1-1.5 hours, and recalibration will only be performed in case of significant signal abnormalities.

SUMMARY:
Non-invasive ventilation (NIV) has been widely used in heart failure patients with supporting evidence. However, the drawbacks and contraindications associated with NIV limit its applicability in certain patients. Recently, high-flow oxygen therapy (HFOT) has gained popularity, particularly in the context of the COVID-19 pandemic, due to its documented benefits, improved patient comfort and fewer contraindications. Studies have suggested that HFOT can generate positive end-expiratory pressure (PEEP) similar to NIV, thereby increasing end-expiratory lung volume. However, the specific effects of PEEP remain unknown, as previous research only monitored the upper airway pressure. Therefore, this study aims to explore the flow-pressure relationship between HFOT and NIV in heart failure patients using electrical impedance tomography (EIT).

This prospective randomized crossover clinical trial will be conducted at a single medical center with multiple intensive care units. Participants will be randomly assigned to Groups A and B using a computerized randomization process. Each group will undergo specific protocols for 5-10 minutes per phase, during which parameters including respiratory rate, heart rate, blood pressure, peripheral oxygen saturation, and oxygen concentration will be recorded. NIV will be administered in continuous positive airway pressure (CPAP) mode. Additional parameters such as tidal volume, respiratory rate, minute ventilation, leak flow, and peak inspiratory pressure will be recorded for NIV.

The study protocols for Group A will follow the sequence of oxygen mask, HFOT 40L, HFOT 50L, HFOT 60L, oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, and CPAP 6cmH2O. Group B will follow the sequence of oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, CPAP 6cmH2O, oxygen mask, HFOT 40L, HFOT 50L, and HFOT 60L. This means that each intervention will be performed in the order listed, with one intervention completed before moving on to the next.

The participants will be positioned in a semi-recumbent position at 45 degrees, and the EIT belt will be placed around the fifth (or sixth) intercostal space for monitoring. The EIT signals will be filtered with a cut-off frequency set at 10 beats below the current heart rate. The entire procedure is estimated to take approximately 1-1.5 hours, and recalibration will only be performed in case of significant signal abnormalities. All data will be stored for offline analysis.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) has been widely used in heart failure patients with supporting evidence. However, the drawbacks and contraindications associated with NIV limit its applicability in certain patients. Recently, high-flow oxygen therapy (HFOT) has gained popularity, particularly in the context of the COVID-19 pandemic, due to its documented benefits, improved patient comfort and fewer contraindications. Studies have suggested that HFOT can generate positive end-expiratory pressure (PEEP) similar to NIV, thereby increasing end-expiratory lung volume. However, the specific effects of PEEP remain unknown, as previous research only monitored the upper airway pressure. Therefore, this study aims to explore the flow-pressure relationship between HFOT and NIV in heart failure patients using electrical impedance tomography (EIT).

This prospective randomized crossover clinical trial will be conducted at a single medical center with multiple intensive care units. Participants will be randomly assigned to Groups A and B using a computerized randomization process. Each group will undergo specific protocols for 5-10 minutes per phase, during which parameters including respiratory rate, heart rate, blood pressure, peripheral oxygen saturation, and oxygen concentration will be recorded. NIV will be administered in continuous positive airway pressure (CPAP) mode. Additional parameters such as tidal volume, respiratory rate, minute ventilation, leak flow, and peak inspiratory pressure will be recorded for NIV.

The study protocols for Group A will follow the sequence of oxygen mask, HFOT 40L, HFOT 50L, HFOT 60L, oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, and CPAP 6cmH2O. Group B will follow the sequence of oxygen mask, CPAP 4cmH2O, CPAP 5cmH2O, CPAP 6cmH2O, oxygen mask, HFOT 40L, HFOT 50L, and HFOT 60L. This means that each intervention will be performed in the order listed, with one intervention completed before moving on to the next.

The participants will be positioned in a semi-recumbent position at 45 degrees, and the EIT belt will be placed around the fifth (or sixth) intercostal space for monitoring. The EIT signals will be filtered with a cut-off frequency set at 10 beats below the current heart rate. The entire procedure is estimated to take approximately 1-1.5 hours, and recalibration will only be performed in case of significant signal abnormalities. All data will be stored for offline analysis.

The primary outcome will compare the difference of global end-expiratory lung impedance (ΔEELI) between HFOT with a flow rate of 40 L/min and NIV with CPAP 4 cmH2O. The secondary study aims to assess the corresponding PEEP values in NIV with CPAP under different airflow rates during HFOT.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the intensive care unit (ICU) with PaO2/FiO2 ≤ 300, requiring Non-Invasive Ventilation (NIV) and High-Flow Oxygen Therapy (HFOT) and stable use of NIV and HFOT for at least 24 hours will be eligible for enrollment.
* Evidence of pulmonary infiltrates on chest X-ray in patients with heart failure.
* Alert and able to follow instructions.

Exclusion Criteria:

* Age < 18 years.
* Patients with a history of tracheostomy.
* Hemodynamically unstable (defined as a mean arterial pressure persistently below 60 mmHg despite fluid resuscitation or vasopressor support).
* Severe chronic obstructive pulmonary disease (COPD).
* History of nasal trauma and/or nasal septal deviation or any other reason preventing the use of High-Flow Oxygen Therapy (HFOT).
* Presence of facial wounds or any other reason preventing the use of Non-Invasive Ventilation (NIV).
* Contraindications to Electrical Impedance Tomography (EIT) use (e.g., patients with implanted pacemakers) or inability to place EIT belt (e.g., due to wound dressings or chest drainage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
compare the difference of global end-expiratory lung impedance (ΔEELI) between HFOT and NIV | approximately 1-1.5 hours
  compare the difference of global end-expiratory lung impedance (ΔEELI) between HFOT with a flow rate of 40 L/min and NIV with CPAP 4 cmH2O.

SECONDARY OUTCOMES:
PEEP values in NIV with CPAP under different airflow rates during HFOT | approximately 1-1.5 hours
  assess the ΔEELI corresponding PEEP values in NIV with CPAP under different airflow rates during HFOT

CONTACTS AND LOCATIONS:
Overall Officials: MING-HANN SHIN, Principal Investigator — Division of Respiratory Therapy, Department of Integrated Diagnostic and Therapeutics, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Background] Plotnikow GA, Thille AW, Vasquez DN, Pratto RA, Quiroga CM, Andrich ME, Dorado JH, Gomez RS, D'Annunzio PA, Scapellato JL, Intile D. Effects of High-Flow Nasal Cannula on End-Expiratory Lung Impedance in Semi-Seated Healthy Subjects. Respir Care. 2018 Aug;63(8):1016-1023. doi: 10.4187/respcare.06031. Epub 2018 Jun 26. PMID 29945910
- [Background] Yuan Z, Han X, Wang L, Xue P, Sun Y, Frerichs I, Moller K, Xing J, Zhao Z. Oxygen Therapy Delivery and Body Position Effects Measured With Electrical Impedance Tomography. Respir Care. 2020 Mar;65(3):281-287. doi: 10.4187/respcare.07109. Epub 2019 Nov 26. PMID 31772064
- [Result] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Result] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Result] Nielsen KR, Ellington LE, Gray AJ, Stanberry LI, Smith LS, DiBlasi RM. Effect of High-Flow Nasal Cannula on Expiratory Pressure and Ventilation in Infant, Pediatric, and Adult Models. Respir Care. 2018 Feb;63(2):147-157. doi: 10.4187/respcare.05728. Epub 2017 Oct 24. PMID 29066588
- [Result] Zhang R, He H, Yun L, Zhou X, Wang X, Chi Y, Yuan S, Zhao Z. Effect of postextubation high-flow nasal cannula therapy on lung recruitment and overdistension in high-risk patient. Crit Care. 2020 Mar 6;24(1):82. doi: 10.1186/s13054-020-2809-7. PMID 32143664
- [Result] Perez-Teran P, Marin-Corral J, Dot I, Sans S, Munoz-Bermudez R, Bosch R, Vila C, Masclans JR. Aeration changes induced by high flow nasal cannula are more homogeneous than those generated by non-invasive ventilation in healthy subjects. J Crit Care. 2019 Oct;53:186-192. doi: 10.1016/j.jcrc.2019.06.009. Epub 2019 Jun 19. PMID 31254850